CLINICAL TRIAL: NCT06344039
Title: Epidemiological Study of Floating Hip Injuries in Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Yaser Emam Mohamed, Resident Doctor, Assiut University
Other Study IDs: Floating hip
Record Dates: First submitted 2024-03-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hip Fractures; Hip Injuries
Keywords: Floating hip; Pelvic fractures; Acetabular fractures; Femur fractures; Trauma
MeSH Terms: conditions — Hip Fractures; Hip Injuries; Femoral Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is to describe and study the patterns of floating hip injuries and assess the current management in Assiut University Hospitals Trauma Centre to help reach the best approach to plan treatment for these severe and difficult injuries.

DETAILED DESCRIPTION:
Floating hip injuries are defined as ipsilateral fractures of the pelvis, acetabulum and femur . The term "floating" is used in orthopedic literature to describe certain patterns of skeletal injuries that share one common character which is disruption and discontinuity of bones above and below a joint. This type of injury is very rare and occurs due to high-energy trauma most commonly road traffic accidents and falls from height. Patients of the floating hip injuries are usually poly-trauma patients with other associated potentially serious injuries in the head , chest or abdomen or fractures in other sites. Complication rates are high in these patients due to the severe and unstable nature of this injury. The femoral fracture may be associated with pelvic, acetabular fracture or both, this pattern was classified by Liebergall et al into 3 types; A, B and C with type A involving pelvic fracture associated with an ipsilateral femoral fracture and type B involving an acetabular fracture associated with an ipsilateral femoral fracture and type C involving fractures to both the pelvis and acetabulum. The lack of common terminology , probably because of their rarity and relative low incidence of associated vascular injuries , could have been the reason for the underappreciation of the peculiarity of these injuries. Previous studies have been limited in number without deep analysis of the current practice patters and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 to 60) with ipsilateral fractures of the pelvis, acetabulum and femur

Exclusion Criteria:

* Ages below 18 or above 60
* pathological and fragility fractures

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All patients aged 18 to 60 who were admitted to Assiut University Hospitals and presented with ipsilateral fractures of the pelvis, acetabulum, and femur in the period between 2018-2023
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of floating hip injuries | From 2018-2023
  Determination of the incidence rate of injury by calculating new cases / total number of trauma cases admitted in the time frame from 2018-2023
Patterns of injury | 2018-2023
  Determination of patterns of injury using the liebergall classification . Fractures are classified into A, B, and C and their percentages over the total number of cases will be calculated

REFERENCES:
- [Background] Yang Y, Zou C, Fang Y, Shakya S. Medium-term clinical results in patients with floating hip injuries. BMC Surg. 2023 Feb 20;23(1):40. doi: 10.1186/s12893-023-01927-6. PMID 36803387
- [Background] Muller EJ, Siebenrock K, Ekkernkamp A, Ganz R, Muhr G. Ipsilateral fractures of the pelvis and the femur--floating hip? A retrospective analysis of 42 cases. Arch Orthop Trauma Surg. 1999;119(3-4):179-82. doi: 10.1007/s004020050385. PMID 10392514
- [Background] Liebergall M, Mosheiff R, Safran O, Peyser A, Segal D. The floating hip injury: patterns of injury. Injury. 2002 Oct;33(8):717-22. doi: 10.1016/s0020-1383(01)00204-2. PMID 12213424
- [Background] Wu CL, Tseng IC, Huang JW, Yu YH, Su CY, Wu CC. Unstable pelvic fractures associated with femoral shaft fractures: a retrospective analysis. Biomed J. 2013 Mar-Apr;36(2):77-83. doi: 10.4103/2319-4170.110401. PMID 23644236
- [Background] Zamora-Navas P, Guerado E. Vascular complications in floating hip. Hip Int. 2010;20 Suppl 7:S11-8. doi: 10.1177/11207000100200s703. Epub 2010 May 27. PMID 20512766
- [Background] Mohamed SO, Ju W, Qin Y, Qi B. The term "floating" used in traumatic orthopedics. Medicine (Baltimore). 2019 Feb;98(7):e14497. doi: 10.1097/MD.0000000000014497. PMID 30762776
- [Background] Burd TA, Hughes MS, Anglen JO. The floating hip: complications and outcomes. J Trauma. 2008 Feb;64(2):442-8. doi: 10.1097/TA.0b013e31815eba69. PMID 18301213
- [Background] Brioschi M, Randelli F, Capitani P, Capitani D. Floating hip in polytraumatized patients: complications, mechanism of injury, and surgical strategy. Int Orthop. 2022 Feb;46(2):361-368. doi: 10.1007/s00264-021-05262-4. Epub 2021 Nov 15. PMID 34779899
- [Background] Meena UK, Bansal MC, Behera P, Goyal D, Kumar R. Concomitant ipsilateral acetabular and femoral fractures - an appraisal of outcomes and complications in 34 patients. Acta Orthop Belg. 2021 Sep;87(3):401-410. PMID 34808712
- [Background] Cech A, Rieussec C, Kerschbaumer G, Seurat O, Corbet C, Vibert B, Tronc C, Ruatti S, Bouzat P, Tonetti J, Boudissa M. Complications and outcomes in 69 consecutive patients with floating hip. Orthop Traumatol Surg Res. 2021 Oct;107(6):102998. doi: 10.1016/j.otsr.2021.102998. Epub 2021 Jun 29. PMID 34214653
- [Background] Liebergall M, Lowe J, Whitelaw GP, Wetzler MJ, Segal D. The floating hip. Ipsilateral pelvic and femoral fractures. J Bone Joint Surg Br. 1992 Jan;74(1):93-100. doi: 10.1302/0301-620X.74B1.1732275.